CLINICAL TRIAL: NCT06400914
Title: Clinical Evaluation of Biomedics Monthly Sphere and Avaira Vitality Sphere
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Collaborators: Centre for Ocular Research & Education, Canada (Other)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EX-MKTG-156
Record Dates: First submitted 2024-04-24; First posted 2024-05-06 (Actual); Results first posted 2025-07-03 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Ametropia
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Lens A (ocufilcon D) (Experimental): All participants will wear lens A for 15 minutes (Period 1).
  Interventions: Device: Lens A (ocufilcon D)
- Lens B (fanfilcon A) (Experimental): All participants will wear lens B for 15 minutes (Period 2).
  Interventions: Device: Lens B (fanfilcon A)

INTERVENTIONS:
Device: Lens A (ocufilcon D) — 15 minutes of daily wear.
  Arms: Lens A (ocufilcon D)
Device: Lens B (fanfilcon A) — 15 minutes of daily wear.
  Arms: Lens B (fanfilcon A)

SUMMARY:
The aim of this study is to compare the short-term clinical performance of two sphere contact lenses.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the short-term clinical performance of two different sphere contact lenses after 15 minutes of daily wear each.

ELIGIBILITY:
Inclusion Criteria:

1. Is at least 18 years of age and has full legal capacity to volunteer.
2. Has read and signed an information consent letter.
3. Self-reports having a full eye examination in the previous two years.
4. Anticipates being able to wear the study lenses for the required time of the study.
5. Is willing and able to follow instructions and maintain the appointment schedule.
6. Has refractive astigmatism no higher than -0.75 DC.
7. Can be fit with the available lens parameters (sphere +6.00 to -10.00D).
8. Can achieve binocular distance vision of at least 20/30 Snellen (logMAR 0.18) with the study contact lenses.

Exclusion Criteria:

1. Is participating in any concurrent clinical or research study.
2. Has any known active ocular disease and/or infection that contraindicates contact lens wear.
3. Has a systemic condition that in the opinion of the investigator may affect a study outcome variable.
4. Is using any systemic or topical medications that in the opinion of the investigator may affect contact lens wear or a study outcome variable.
5. Has known sensitivity to the diagnostic sodium fluorescein used in the study.
6. Self-reports as pregnant, lactating or planning a pregnancy at the time of enrolment.
7. Has undergone refractive error surgery or intraocular surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-04-03 (Actual); Primary Completion 2024-05-11 (Actual); Study Completion 2024-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Guerrero, MSc, FIACLE, Principal Investigator — National Autonomous University
Locations (1):
- Consultorio Optométrico Queretaro, Mexico City, Mexico

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Forty-four participants were screened and dispensed lenses. All participants who were dispensed with lenses completed the study. (n=44)
Groups:
- Lens A (Ocufilcon D): All participants wore lens A for 15 minutes (Period 1).
  Lens A (ocufilcon D): 15 minutes of daily wear.
- Lens B (Fanfilcon A): All participants wore lens B for 15 minutes (Period 2).
  Lens B (fanfilcon A): 15 minutes of daily wear.
Period: Period 1: Lens A (15 Minutes)
Arm/Group | Lens A (Ocufilcon D) | Lens B (Fanfilcon A)
Started | 44 | 0 (All participants received Lens A in Period 1.)
Completed | 44 | 0
Not Completed | 0 | 0
Period: Period 2: Lens B (15 Minutes)
Arm/Group | Lens A (Ocufilcon D) | Lens B (Fanfilcon A)
Started | 0 (All participants received Lens B in Period 2.) | 44
Completed | 0 | 44
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Includes all study participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.7 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Lens Fit Acceptance Ratings
Description: Overall lens fit acceptance was measured on a scale from 0-4 (0=Should not be worn and 4= Perfect)
Time Frame: At the end of 15 Minutes of wear
Population: All the forty-four participants who started the study, completed the study.
Measure: Mean (Standard Deviation); unit: Units on Scale
Arm/Group | Lens A (Ocufilcon D) | Lens B (Fanfilcon A)
Number analyzed (Participants) | 44 | 44
Units on Scale | 3.3 (1.1) | 3.7 (0.8)

ADVERSE EVENTS:
Time Frame: Through study completion, approximately five weeks.
Arm/Group | Lens A (Ocufilcon D) | Lens B (Fanfilcon A)
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 0/44 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-06): https://cdn.clinicaltrials.gov/large-docs/14/NCT06400914/Prot_SAP_000.pdf